CLINICAL TRIAL: NCT06481683
Title: Evaluation of Maternal Serum Stathmin-1 Levels as a Biomarker in Preeclampsia and Severe Preeclampsia
Brief Title: Maternal Serum Stathmin-1 Levels in Preeclampsia
Acronym: MSSLP
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to the change of the clinic where the principal investigator was employed.
Sponsor: Burak Yücel Special Clinic (Other)
Responsible Party: Principal Investigator, Burak Yücel, Dr., Burak Yücel Special Clinic
Other Study IDs: Stathmin_2022.08.275
Record Dates: First submitted 2024-06-24; First posted 2024-07-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Preeclampsia
Keywords: Stathmin-1; Preeclampsia; Severe Preeclampsia; Trophoblast invasion; Maternal serum biomarkers
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-eclampsia Group (Case Group): This group consists of pregnant women diagnosed with pre-eclampsia. These participants will have specific characteristics related to the pre-eclampsia condition, such as elevated blood pressure and proteinuria.
- Severe Pre-eclampsia Group (Case Group): This group consists of pregnant women diagnosed with severe pre-eclampsia. These participants will have more severe symptoms and complications related to pre-eclampsia, potentially including higher blood pressure, significant proteinuria, and other related health issues.
- Control Group: This group consists of pregnant women who do not have pre-eclampsia or severe pre-eclampsia. These participants will be matched to the case groups based on relevant characteristics such as age, gestational age, and other demographic factors.

SUMMARY:
The goal of this observational study is to investigate maternal serum Stathmin-1 levels in pregnancies affected by preeclampsia compared to healthy gestations.

The main questions it aims to answer are:

1. What are the maternal serum Stathmin-1 levels in pregnancies with preeclampsia?
2. How do Stathmin-1 levels differ between preeclampsia with severe features and uncomplicated pregnancies?

Researchers will compare Stathmin-1 levels in pregnancies with preeclampsia and preeclampsia with severe features to those in a control group of healthy pregnancies to assess differences in biomarker levels.

Participants will undergo blood sample collection at 32-34 weeks of gestation. Have their blood samples processed for Stathmin-1 level measurement using ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age: Pregnancies between 20 weeks and term (up to 40 weeks).
* Diagnosis of Preeclampsia (PE): New-onset hypertension (systolic BP ≥140 mmHg and/or diastolic BP ≥90 mmHg) after 20 weeks of gestation, with or without proteinuria.
* Diagnosis of Severe Preeclampsia: Defined by criteria such as severe hypertension (systolic BP ≥160 mmHg or diastolic BP ≥110 mmHg), organ dysfunction (renal insufficiency, liver involvement, neurological complications), thrombocytopenia, pulmonary edema, or fetal growth restriction.
* Control Group: Healthy pregnancies without preeclampsia or other significant maternal or fetal complications.

Exclusion Criteria:

* Multiple Pregnancies: Participants carrying more than one fetus.
* Pregestational Diabetes: Pre-existing diabetes mellitus diagnosed before pregnancy.
* Chronic Hypertension: Pre-existing hypertension diagnosed before pregnancy or before 20 weeks of gestation.
* Systemic Diseases: Chronic kidney disease, autoimmune diseases, or other significant systemic illnesses.
* Fetal Anomalies: Identified structural or genetic abnormalities in the fetus.
* Premature Rupture of Membranes: Spontaneous rupture of membranes before the onset of labor at term (37 weeks of gestation) or preterm (before 37 weeks of gestation).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population from which the groups or cohorts in this study will be selected likely consists of pregnant women receiving care at a referral center for maternal care.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Maternal Serum Stathmin-1 Levels | Measured at the time of diagnosis and followed up until delivery.
  To identify and compare Maternal Serum Stathmin-1 Levels levels between the pre-eclampsia group, severe pre-eclampsia group, and the control group. This will help in understanding the biochemical environment associated with pre-eclampsia and its severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No